CLINICAL TRIAL: NCT04264871
Title: Is the Preoperative Preparation of Sickle Cell Patients Optimal: Retrospective Assessment of Practices and Post-operative Complications in a Cohort of Children Followed at Hôpital Universitaire Des Enfants Reine Fabiola (HUDERF) and Who Have Been Managed According Local Guidelines Including Transfusion or Exchange Transfusion Before Surgery
Brief Title: Is the Preoperative Preparation of Sickle Cell Patients Optimal: Assessment of Practices and Post-operative Complications
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Queen Fabiola Children's University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: P2020/Hemato/SCDPreop
Record Dates: First submitted 2020-02-07; First posted 2020-02-11 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-01

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Children with sickle cell disease systematically receive a transfusion 2 to 5 days before scheduled surgery (with the exception of minor surgeries) in order to avoid post-operative complications of which the vaso-occlusive crisis and acute thoracic syndrome are the most frequent.

This standardized preoperative protocol was established on the basis of the results of large-scale randomized studies, most of which date back over ten years, and which have demonstrated the beneficial effects of transfusion (or transfusion exchange) preoperatively. To date, several other more recent studies (but not controlled) have questioned this type of systematic management.

The purpose of this study is to review retrospectively data of sickle cell children who have undergone elective surgery at the Huderf in the last ten years and to identify the eventual complications encountered. The most common procedures in these patients are: tonsillectomy with or without associated adenoids, splenectomy and cholecystectomy.

General data on sickle cell disease (history, genotype, G6PD deficiency, biology and previous complications), pre-surgical preparation, surgery and post surgical management and complications will be collected and analyzed.

This retrospective analysis will allow an objective assessment of the current quality of care and will provide useful data to improve patient management.

ELIGIBILITY:
Inclusion Criteria:

* Sickle cell disease with surgery during the 2010-2019 period

Exclusion Criteria:

* None

Max Age: 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients with sickle cell disease followed at Hôpital Universitaire des Enfants Reine Fabiola and having undergone a surgery betwee 2010-2019
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-05-31 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
To assess the overall incidence of vaso-occlusive-events 1 month post surgery | 1 month after surgery
  Vaso-occlusive-events will include Vaso Occlusive Crisis (acute pain events that requires a visit to a medical facility and administration of pain medications (opioids or IV NSAIDs)), acute chest syndrome (new pulmonary infiltrate associated with by pneumonia-like symptoms, pain or fever) and hemoglobin < 6g/dl

SECONDARY OUTCOMES:
To assess the incidence of Vaso Occlusive Crisis 1 month post surgery | 1 month after surgery
  Vaso Occlusive Crisis is defined as acute pain events that requires a visit to a medical facility and administration of pain medications (opioids or IV NSAIDs)
To assess the incidence of Vaso Occlusive Crisis 3 months post surgery | 3 months after surgery
  Vaso Occlusive Crisis is defined as acute pain events that requires a visit to a medical facility and administration of pain medications (opioids or IV NSAIDs)
To assess the incidence of Vaso Occlusive Crisis 12 months post surgery | 12 months after surgery
  Vaso Occlusive Crisis is defined as acute pain events that requires a visit to a medical facility and administration of pain medications (opioids or IV NSAIDs)
To assess the incidence of Acute Chest Syndrome 1 month post surgery | 1 month after surgery
  Acute Chest Syndrome is defined as a new pulmonary infiltrate associated with by pneumonia-like symptoms, pain or fever
To assess the incidence of Acute Chest Syndrome 3 months post surgery | 3 months after surgery
  Acute Chest Syndrome is defined as a new pulmonary infiltrate associated with by pneumonia-like symptoms, pain or fever
To assess the incidence of Acute Chest Syndrome 12 months post surgery | 12 months after surgery
  Acute Chest Syndrome is defined as a new pulmonary infiltrate associated with by pneumonia-like symptoms, pain or fever
To assess the duration of hospitalization post-surgery | 1 month after surgery
  number of days between surgery and day of discharge
To assess the incidence of Red Blood Cell (RBC) allo-immunization 1 month post surgery | 1 month after surgery
  incidence of acute anemia with the presence of new allo-antibody(ies) against RBC
To assess the incidence of RBC allo-immunization 3 months post surgery | 3 months after surgery
  incidence of acute anemia with the presence of new allo-antibody(ies) against RBC
To assess the incidence of RBC allo-immunization 12 months post surgery | 12 months after surgery
  incidence of acute anemia with the presence of new allo-antibody(ies) against RBC
To assess the number of RBC transfusion episodes 1 month post surgery | 1 month after surgery
  Number of RBC unit transfused

CONTACTS AND LOCATIONS:
Overall Officials: Alina Ferster, MD, Principal Investigator — Queen Fabiola Children's University Hospital
Locations (1):
- Hôpital Universitaire Des Enfants Reine Fabiola, Brussels, Brussles, Belgium